CLINICAL TRIAL: NCT07149883
Title: Evaluation of Mean Platelet Volume and Systemic Inflammatory Response Index (SIRI) in Patients of Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa salama ahmed omar, Doctor, Assiut University
Other Study IDs: MPV and SIRI in of ACS
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Complete blood count — Complete blood count
Device: ECHO — device that used to evaluate the cardiac function

SUMMARY:
To assess the diagnostic and prognostic significance of MPV and SIRI in patients presenting with acute coronary syndrome.(STEMI/NSTEMI/UN STABLE ANGINA)

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS), which includes unstable angina, non-ST elevation myocardial infarction (NSTEMI), and ST elevation myocardial infarction (STEMI), is a leading cause of hospitalization and death globally【1】. The pathophysiology of ACS involves plaque rupture, platelet activation, thrombus formation, and a significant inflammatory component【2】. Early diagnosis and accurate risk stratification are critical for improving patient outcomes and guiding therapy.

Mean Platelet Volume (MPV) is a simple, cost-effective parameter obtained from the complete blood count. It reflects platelet size and activity-larger platelets are more reactive and thrombogenic. Studies have demonstrated that MPV is elevated in patients with ACS and may correlate with infarct size and poor prognosis【3,4】.

The systemic inflammatory response plays a pivotal role in the destabilization of atherosclerotic plaques. Recently, novel inflammatory indices such as the Systemic Inflammatory Response Index (SIRI)-calculated as (neutrophil count × monocyte count) / lymphocyte count-have emerged as potential marker for cardiovascular risk. SIRI reflects the combined effect of pro-inflammatory and anti-inflammatory components of the immune system【5】. Elevated SIRI has been associated with adverse outcomes in various conditions, including stroke, cancer, and cardiovascular diseases【6,7】.

Despite the individual significance of MPV and SIRI, limited data are available on their combined utility in ACS patients. Evaluating both markers together may provide a more comprehensive picture of the thrombo-inflammatory state and help identify high-risk patients at admission, facilitating more personalized care【8】.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.

  * Diagnosed with acute coronary syndrome (unstable angina, NSTEMI, STEMI).
  * Admission within 24 hours of symptom onset.

Exclusion Criteria:

* o Active infection or chronic inflammatory diseases.

  * Known hematological disorders or malignancy.
  * Chronic liver or renal failure.
  * Recent surgery or trauma (< 1 month).
  * Patients with rheumatic heart disease
  * Patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute coronary syndrome (ACS), which includes unstable angina, non-ST elevation myocardial infarction (NSTEMI), and ST elevation myocardial infarction (STEMI), is a leading cause of hospitalization and death globally【1】. The pathophysiology of ACS involves plaque rupture, platelet activation, thrombus formation, and a significant inflammatory component【2】. Early diagnosis and accurate risk stratification are critical for improving patient outcomes and guiding therapy.
  Mean Platelet Volume (MPV) is a simple, cost-effective parameter obtained from the complete blood count. It reflects platelet size and activity-larger platelets are more reactive and thrombogenic. Studies have demonstrated that MPV is elevated in patients with ACS and may correlate with infarct size and poor prognosis【3,4】.
  The systemic inflammatory response plays a pivotal role in the destabilization of atherosclerotic plaques. Recently, novel inflammatory indices such as the Systemic Inflammatory Response Index (SIRI)-
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic and prognostic significance of MPV and SIRI in patients presenting with acute coronary syndrome.(STEMI/NSTEMI/UN STABLE ANGINA) | Baseline
  Evaluation of mean platelet volume and systemic inflammatory response index (SIRI) in patients of acute coronary syndrome

SECONDARY OUTCOMES:
To assess the diagnostic and prognostic significance of MPV and SIRI in patients presenting with acute coronary syndrome.(STEMI/NSTEMI/UN STABLE ANGINA | Baseline
  Evaluation of mean platelet volume and systemic inflammatory response index (SIRI) in patients of acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Hassan, Professor, Study Director — Assuit university hospital; Hanan Sharaf, Professor, Study Director — Assuit university hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Libby P. Inflammation in atherosclerosis. Nature. 2002 Dec 19-26;420(6917):868-74. doi: 10.1038/nature01323. PMID 12490960
- [Background] Anderson JL, Morrow DA. Acute Myocardial Infarction. N Engl J Med. 2017 May 25;376(21):2053-2064. doi: 10.1056/NEJMra1606915. No abstract available. PMID 28538121